CLINICAL TRIAL: NCT03202537
Title: Effectiveness of Physiologic Testing in PPI Non-Responders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Washington University School of Medicine (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Pandolfino, Professor of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00204123
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dexlansoprazole (Experimental): dexlansoprazole 90mg per day (60mg am, 30mg pm dosing) for 4 weeks
  Interventions: Drug: dexlansoprazole

INTERVENTIONS:
Drug: dexlansoprazole — dexlansoprazole treatment for Gastroesophageal Reflux symptoms
  Other Names: Dexilant

SUMMARY:
The prevalence of GERD is estimated to be as high as 20% in the US, and up to 50% remain symptomatic on proton pump inhibitor (PPI) therapy. The clinical approach to understand the mechanism of nonresponse is not standardized, and patients will often undergo various tests: 1) pH-impedance, 2) wireless pH monitoring over 96 hours, 3) high-resolution impedance manometry (HRIM), and 4) mucosal impedance (MI). Controversy exists regarding the best technique, optimal study protocol and treatment approach for the PPI non-responder (PPINR) group, resulting in inappropriate resource utilization and a failure to provide effective personalized care. The first aim is to identify the relevant physiologic parameters of diagnostic tools in their ability to predict PPI requirement. In Aim Two, these results will be applied to guide the formal development of a clinical algorithm for the management of PPINRs with personalized clinical pathways based on mechanism of treatment failure. We will first perform a prospective comparison trial of 240 PPINR subjects at 2 sites over 4 years. Subjects will complete symptom questionnaires and undergo diagnostic testing (pH-impedance on PPI therapy, HRIM, 96-hr wireless pH monitoring off PPI therapy and MI). Those who have a positive pH study and/or resume PPI therapy will receive escalation of therapy with dexlansoprazole. We will compare the ability of 96-hr wireless pH monitoring vs pH impedance to predict PPI requirement and response to dexlansoprazole, respectively. We will explore whether MI is equivalent to 96-hr wireless pH monitoring in predicting PPI requirement. Lastly, we will determine whether HRIM metrics can be utilized to determine reflux burden, mechanism and response to treatment. Next, the investigators will develop quality measures for reflux testing in order to develop a simplified management strategy for the PPINR group. The RAND/UCLA Appropriateness Methodology will be utilized with an expert working group to develop formal validated quality measures for reflux testing.

DETAILED DESCRIPTION:
The prevalence of gastroesophageal reflux disease is estimated to be as high as 20% in the United States, and up to 50% of these patients remain symptomatic on proton pump inhibitor (PPI) therapy. Unfortunately, the clinical approach to understand the mechanism of nonresponse is not standardized, and patients will often undergo various esophageal function tests: 1) pH-impedance, 2) wireless pH monitoring over 96 hours, 3) high-resolution impedance manometry (HRIM), and 4) mucosal impedance. Currently significant controversy exists regarding the best technique, optimal study protocol and treatment approach for the PPI non-responder (PPINR) group, resulting in inappropriate resource utilization and a failure to provide effective personalized care. As such, PPINRs contribute to a large healthcare burden in the United States.

The first aim of the study is to identify the relevant physiologic parameters of the aforementioned diagnostic tools in their ability to predict PPI requirement. Subsequently, in Aim Two, these results will be applied to guide the formal development of a clinical algorithm for the management of PPINRs with personalized clinical pathways based on mechanism of treatment failure.

The investigators will first perform a prospective comparison trial of 240 PPINR subjects at two centers over a 4 year period. Subjects will complete symptom questionnaires and undergo diagnostic testing (pH-impedance on PPI therapy, HRIM, 96-hthe wireless pH monitoring off of PPI therapy and mucosal impedance). Those who have a positive pH study and/or resume PPI therapy will receive escalation of acid suppression therapy with dexlansoprazole. Experiments 1a & 1b will compare the ability of 96-hthe wireless pH monitoring vs pH impedance to predict PPI requirement and response to dexlansoprazole, respectively. Experiment 1c will explore whether mucosal impedance is equivalent to 96-hthe wireless pH monitoring in predicting PPI requirement. Lastly, Experiment 1d will determine whether HRIM metrics can be utilized to determine reflux burden, mechanism and response to treatment. Next, the investigators will develop quality measures for reflux testing in order to develop a simplified management strategy for the PPINR group. The RAND/UCLA Appropriateness Methodology will be utilized with an expert working group to develop formal validated quality measures for reflux testing based on results from aim 1 in addition to the available literature & evidence. This will be conducted over twelve months (years 4 to 5).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-80 years old (females of childbearing potential should be on highly effective contraceptive methods)
* Mentally capable to provide informed consent in English
* Present to the Northwestern Medical Group GI practice or the Washington University Division of Gastroenterology with symptoms of GERD (heartburn, regurgitation, and non-cardiac chest pain)
* Have failed an appropriate compliant trial of PPI therapy with a GERD-Q score ≥8.
* Able to undergo endoscopy, ambulatory reflux monitoring, manometry, PPI therapy cessation and trial of dexlansoprazole therapy. Subjects with Los Angeles Classification Grade A (mild) or B esophagitis and symptomatic, non-erosive disease will be enrolled.

Exclusion Criteria:

* Participation in a concurrent clinical trial or completed another trial within past 8 weeks.
* Active severe erosive esophagitis (Los Angeles Grade C or D), long-segment Barrett's esophagus (Zap score of 4)
* Eosinophilic esophagitis
* Prior gastrointestinal surgery of the esophagus and/or stomach
* Current treatment with dexlansoprazole
* Current signs or symptoms of heart disease. All patients with non-cardiac chest pain are required to have a cardiologist evaluation as standard of care work up in the evaluation of non-cardiac chest pain.
* Subjects with clinically abnormal results of the screening ECG and/or chemistry panel (particularly prolonged QTc interval or hypomagnesaemia) excluded from the dexlansoprazole trial. Subjects with sensitivities or allergies to the metals contained in the Bravo capsule including chromium, nickel, copper, cobalt, and iron.
* Unstable medical illness with ongoing diagnostic work-up and treatment. Patients with well-controlled hypertension, diabetes and a remote history of ischemic heart disease that is deemed stable, as judged by the investigator can be included.
* History of drug addiction, drug abuse or alcoholism.
* Current neurologic or cognitive impairment, which would preclude ability to obtain informed consent.
* Pregnant patients.
* Patients with Cirrhosis (Childs Classification A-C).Special vulnerable populations including children, prisoners, institutionalized individuals.
* Bleeding disorder or requirement of NSAID/aspirin during monitoring period.
* Drugs that affect gastrointestinal symptoms (H2 blockers, antacids, metoclopramide, domperidone, erythromycin, anticholinergics [bentyl, levsin, belladonna etc.]). Antidepressants can be continued at stable dose.
* Drugs listed on the Dexilant label including antiretrovirals (Rilpivirine-containing products, Atazanavir, Nelfinavir, Saquinavir, etc), Warfarin, Methotrexate, Drugs Dependent on Gastric pH for Absorption (e.g., iron salts, erlotinib, dasatinib, nilotinib, mycophenolate mofetil, ketoconazole/itraconazole), Tacrolimus, CYP2C19 or CYP3A4 Inducers or inhibitors.
* Patients found to have achalasia, a spastic disorder, hypercontractile disorder or functional obstruction at the esophagogastric junction will be excluded. Subjects with a history of structuring or narrowing upon endoscopy (Subjects with no such history will be enrolled; however, if such features are noted upon endoscopy during the study, these subjects will not undergo MI testing).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
number of patients able to successfully withdraw from PPI treatment | 4.5 years
  ability of 96 hour pH wireless vs pH impedance to predict PPI requirement

CONTACTS AND LOCATIONS:
Overall Officials: John Pandolfino, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Health Care, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyawali CP, Rogers BD, Yadlapati R, Roman S, Carlson DA, Pandolfino J. pH Impedance Monitoring on Proton Pump Inhibitor Therapy Impacts Management Decisions in Proven GERD but Not in Unproven GERD. Clin Gastroenterol Hepatol. 2025 Dec;23(13):2459-2467. doi: 10.1016/j.cgh.2025.02.032. Epub 2025 May 16. PMID 40383216
- [Derived] Yadlapati R, Gyawali CP, Masihi M, Carlson DA, Kahrilas PJ, Nix BD, Jain A, Triggs JR, Vaezi MF, Kia L, Kaizer A, Pandolfino JE. Optimal Wireless Reflux Monitoring Metrics to Predict Discontinuation of Proton Pump Inhibitor Therapy. Am J Gastroenterol. 2022 Oct 1;117(10):1573-1582. doi: 10.14309/ajg.0000000000001871. Epub 2022 Jun 10. PMID 35973148
- [Derived] Yadlapati R, Masihi M, Gyawali CP, Carlson DA, Kahrilas PJ, Nix BD, Jain A, Triggs JR, Vaezi MF, Kia L, Kaizer A, Pandolfino JE. Ambulatory Reflux Monitoring Guides Proton Pump Inhibitor Discontinuation in Patients With Gastroesophageal Reflux Symptoms: A Clinical Trial. Gastroenterology. 2021 Jan;160(1):174-182.e1. doi: 10.1053/j.gastro.2020.09.013. Epub 2020 Sep 16. PMID 32949568